CLINICAL TRIAL: NCT00807352
Title: The Canadian Triage and Acuity Scale for Children; A Prospective Multi-Center Evaluation.
Acronym: PERC CTAS
Status: Completed | Type: Observational
Sponsor: St. Justine's Hospital (Other)
Collaborators: SickKids Foundation (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Jocelyn Gravel, MD, MSC, CHU Sainte-Justine
Other Study IDs: PERC CTAS; Grant No. XG09-049R
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-07

CONDITIONS: Triage; Pediatrics
Keywords: Triage; Pediatrics; Emergency Department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- level 2: Patients triaged level 2
- level 3: patients triaged level 3
- level 4: patients triaged level 4
- level 5: patients triaged level 5

SUMMARY:
The aim of this study is to evaluate the validity and the reproducibility of the canadian triage and acuity scale when applied by regular nurses for the triage of children in the Emergency Department.

DETAILED DESCRIPTION:
The role of triage in the Emergency Department (ED) is to assign high priority to patients who need urgent care while identifying patients that may be able to wait safely. The Canadian Triage and Acuity Scale (CTAS) is a triage tool constructed from a consensus of experts that is universally used in Canada. Until now, there has been no evaluation of the validity of the tool for children in a clinical context. Also, its inter-rater reproducibility has not been evaluated. The expected implementation of a revised version of the Canadian triage tool in 2008 would be an ideal moment to evaluate its validity and reproducibility. Specific objective: 1. To evaluate the validity of the CTAS for children visiting a pediatric ED and 2. To measure the inter-rater agreement for nurses using the CTAS in these settings.

ELIGIBILITY:
Inclusion Criteria:

* Every patient younger than 18 years old that presents to the ED will be eligible except for those that need to go directly to the resuscitation room (triage level 1)

Exclusion Criteria:

* For ethical reasons, patients that need an immediate treatment will not be recruited in the study.
* Patients for whom an informed consent could not be obtained (example: insurmountable language barriers) will not be included.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All children presenting to a pediatric emergency department
Sampling Method: Non-Probability Sample
Enrollment: 1464 (Actual)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The inter-rater agreement between the two nurses measured by the weighted Kappa score | 15 minutes
The correlation between triage level and the hospitalisation rate | 1 day

SECONDARY OUTCOMES:
The correlation between triage level and admission to the intensive care unit | 1 day
The correlation between triage level and length of stay in the ED after being seen by a physician | 1 day
The correlation between triage level and resources use | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Gravel, MD, Principal Investigator — St. Justine's Hospital
Locations (9):
- Canada (9):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's and Women's Hospital, Vancouver, British Columbia
  - IWK Heath Centre, Halifax, Nova Scotia
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - Centre hospitalier de l'Université Laval, Québec, Quebec

REFERENCES:
- [Background] Gravel J, Gouin S, Manzano S, Arsenault M, Amre D. Interrater agreement between nurses for the Pediatric Canadian Triage and Acuity Scale in a tertiary care center. Acad Emerg Med. 2008 Dec;15(12):1262-7. doi: 10.1111/j.1553-2712.2008.00268.x. Epub 2008 Oct 17. PMID 18945238
- [Derived] Gravel J, Gouin S, Goldman RD, Osmond MH, Fitzpatrick E, Boutis K, Guimont C, Joubert G, Millar K, Curtis S, Sinclair D, Amre D. The Canadian Triage and Acuity Scale for children: a prospective multicenter evaluation. Ann Emerg Med. 2012 Jul;60(1):71-7.e3. doi: 10.1016/j.annemergmed.2011.12.004. Epub 2012 Feb 2. PMID 22305329